CLINICAL TRIAL: NCT07359898
Title: International Multicenter Study of the Navitor/Navitor Vision Transcatheter Aortic Valve Platform (The Intensive Study)
Brief Title: International Multicenter Study of the Navitor/Navitor Vision Transcatheter Aortic Valve Platform
Acronym: Intensive
Status: Recruiting | Type: Observational
Sponsor: IRCCS Policlinico S. Donato (Other)
Collaborators: Meditrial SrL (Industry); Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: INTENSIVE CET 264-2025
Record Dates: First submitted 2025-12-16; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-10

CONDITIONS: Severe Native Aortic Stenosis
Keywords: Aortic Stenosis; TAVI; Navitor; Portico
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- Aortic Stenosis Patients: This Study will enroll subjects of all genders who have symptomatic, severe AS, either in native or in a surgical bioprosthetic valve and are indicated for TAVI implantation. The latter can also be predominantly regurgitant to be suitable for enrolment. Subjects must meet all general eligibility criteria for the TAVI procedure and provide written informed consent prior to sites collecting any clinical data for this Study.
  The operative risk determination of study candidates will be done by the local heart team. The assessment of surgical risk will include the Society of Thoracic Surgeons (STS) Adult Cardiac Surgery Risk Calculator score and/or EuroSCORE II, indices of frailty, and comorbidities not captured by risk calculators, as described below, and current TAVI practice guidelines.

SUMMARY:
INTENSIVE is a prospective, single-arm, multi-center, international, investigator-initiated study of the Navitor/Navitor Vision Transcatheter Aortic Valve (Navitor/Navitor Vision Valve) in patients with symptomatic, severe native aortic stenosis to monitor the outcomes of this valve in a real-world clinical setting.

DETAILED DESCRIPTION:
This comprehensive data collection across 25 interventional centers, aligned with standard clinical care practices, seeks to provide an objective benchmark for current TAVR practice.

The Navitor System include the Navitor Transcatheter Aortic Valve (23 mm, 25 mm, 27 mm, 29 mm, and the 35 mm), FlexNav Delivery System (small and large), and Navitor Loading System (small, large, and LG+). The FlexNav Delivery System (small and large) is commercially available in Europe. The 23 mm, 25 mm, 27 mm, 29 mm, and 35 mm valves and their loading systems are currently CE Marked.

The Navitor Valve maintains several design features of the first-generation Portico Valve including same valve sizes and use range (except for the addition of the 35 mm valve to expand the use range), open stent cell design to provide easy coronary access and blood flow, repositionable with the ability to re-sheath and retrieve, leaflets derived from pericardial bovine tissue, and intra-annular placement of leaflets/cuff within the stent frame for early valve function to maintain hemodynamic stability during implant.

The Study will enroll subjects that, after comprehensive Heart Team evaluation, are scheduled for treatment with the Navitor/Navitor Vision Valve according to standard of care at up to 25 experienced TAVI implant centers across Europe and UK. All sites must either have prior Portico or Navitor/Navitor Vision TAVI system experience. Subjects who provide informed consent for the collection of their clinical data in this Study, will undergo Navitor/Navitor Vision Valve implantation via a transfemoral or alternative access (subclavian or axillary) approach using the site's anesthesia protocol for TAVI procedures.

In the Study, the point of enrollment is defined as informed consent signing, whereas the point of registration is defined as the insertion of the FlexNav Delivery System (loaded with a Navitor/Navitor Vision Valve) into the subject's vasculature (the subject is considered attempted with Navitor/Navitor Vision Valve implantation at this point). Only registered subjects will be included in the analysis.

The endpoints of interest will be defined according to VARC-3 definitions. Subjects participating in the Study will be followed for a total of 5 years with data collected at, baseline, procedure, prior to hospital discharge, and follow-up at 30 days, 12 months and annually thereafter up to 5 years.

The expected duration of enrollment is 12 months, and the total duration of the Study including final data cleaning, reporting, and site close-out is expected to be approximately 6.5 years.

This Study will enroll subjects of all genders who have symptomatic, severe AS, either in native or in a surgical bioprosthetic valve and are indicated for TAVI implantation. The latter can also be predominantly regurgitant to be suitable for enrolment. Subjects must meet all general eligibility criteria for the TAVI procedure and provide written informed consent prior to sites collecting any clinical data for this Study.

The operative risk determination of study candidates will be done by the local heart team. The assessment of surgical risk will include the Society of Thoracic Surgeons (STS) Adult Cardiac Surgery Risk Calculator score and/or EuroSCORE II, indices of frailty, and comorbidities not captured by risk calculators, as described below, and current TAVI practice guidelines. A member of the site's clinical investigation team previously trained to the protocol must evaluate patients for the general eligibility criteria, and if applicable, will enter the patients into the site- specific Pre-Screening Log. A patient who does not satisfy all general eligibility criteria prior to informed consent is considered a screen failure and should not be enrolled in the Study.

Sites will ask patients meeting general inclusion criteria and no general exclusion criteria to sign an Informed Consent form following the established Informed Consent process if they wish to participate in the Study.

A patient is considered enrolled in the Intensive Study from the moment the patient provides written informed consent.

Each subject meeting all general eligibility criteria who is enrolled and receives the Navitor valveshall be followed up until completion of the recommended 5 year follow-up period; however, a subject's participation in any clinical study is voluntary and the subject has the right to withdraw at any time without penalty or loss of benefit. Conceivable reasons for discontinuation may include, but not be limited to, the following:

* Subject death
* Subject undergoes the interventional procedure but exits the operating room without an implanted Navitor Valve; in this case, follow-up is limited to 30 days post-procedure for safety assessment
* After Navitor implantation, subject receives another aortic valve intervention during follow-up (eg, valve in valve intervention, surgical AVR, etc): in this case, follow-up is limited to 30 days after the additional procedure for safety assessment
* Subject voluntary withdrawal
* Subject lost-to follow-up as described below
* Subject's follow-up is terminated Sites must collect and document the reason(s) for subject discontinuation. Investigators must also report this to their respective EC as defined by their institution's procedure(s).

No additional follow-up is required or data recorded from subjects once withdrawn from the Study, except for the status (deceased/alive).

In case of subject withdrawal of consent, the site should make attempts to schedule the subject for a final follow-up visit. At this final follow-up visit, the subject will undergo the following assessments (routine assessments during follow-up visit) and related data will be collected when available:

* Echocardiography to include comprehensive transthoracic echocardiogram, including assessment of aortic valve gradients (mean and peak), areas, indices, degree of regurgitation, cardiac output and cardiac index, left ventricle systolic function (global and segmental)
* Adverse Event assessment

ELIGIBILITY:
Inclusion Criteria:

1. Subject is referred to receive a Navitor/Navitor Vision TAVI according to the local Heart Team. The Heart Team determines the indication to TAVI with Navitor/Navitor Vision before the possible enrolment and independently from the study.
2. Subject is of legal age for consent in the host country.
3. Subject has been informed of the nature of the study, agrees to its provisions and has provided written informed consent as approved by the Ethics Committee (EC) of the respective clinical site.

Exclusion Criteria:

1. Pregnant or nursing subjects
2. Need for emergency surgery for any reason
3. Contraindications to Navitor/Navitor Vision TAVI according to the IFU:

   1. Any sepsis, including active endocarditis
   2. Any evidence of left ventricular or atrial thrombus
   3. Vascular conditions (i.e., stenosis, tortuosity, or severe calcification) that make insertion and endovascular access to the aortic valve impossible
   4. Non-calcified aortic annulus
   5. Any leaflet configuration other than tricuspid
   6. Inability to tolerate antiplatelet/anticoagulant therapy
4. Incapacitated individuals, defined as persons who are mentally ill, mentally handicapped, individuals with severe dementia or individuals without legal authority
5. Individuals who are unable to read or write

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This Study will enroll subjects of all genders who have symptomatic, severe AS, either in native or in a surgical bioprosthetic valve and are indicated for TAVI implantation. The latter can also be predominantly regurgitant to be suitable for enrolment.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-10-11 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2031-10 (Estimated)

PRIMARY OUTCOMES:
All cause Mortality | 12 months
  The primary endpoint is all-cause mortality at 12 months post index Navitor/Navitor Vision implantation procedure

SECONDARY OUTCOMES:
Key Valve Academic Research Consortium (VARC) 3 event definitions | 30 days and 12 months
  Secondary (Descriptive) Endpoints:
  The rate of the following key outcomes for the Study will be assessed as descriptive endpoints:
  1. Composite of all-cause mortality, fatal stroke/stroke with disability, type 3/type 4 bleeding, stage 3/stage 4 acute kidney injury, major vascular complications, or major access- related non-vascular complications at 30 days
  2. Composite of all-cause mortality or all stroke at 12 months
  3. Procedural success defined as successful vascular access, delivery and deployment of the Valve; retrieval of the delivery system and correct positioning of a single Valve in the proper anatomical location and the absence of procedural mortality
  4. Mortality at 30 days and 12 months
  5. Stroke at 30 days and 12 months
  6. Transient ischemic attack (TIA) at 30 days and 12 months
  7. Bleeding
  8. Major vascular complications at 30 days
  9. Major access-related non-vascular complications at 30 days
  10. Major cardiac complications at 30 days
Key Valve Academic Research Consortium (VARC) 3 event definitions | 30 days, 3 and 12 months
  11. Acute kidney injury (stage 4, stage 3, and stage 2) at 30 days 12. Permanent pacemaker insertion at 30 days and 12 months 13. Myocardial infarction at 30 days and 12 months 14. Coronary obstruction requiring intervention at 30 days and 12 months 15. Difference in Coronary arteries' cannulation time pre vs post Navitor/Navitor Vision implant 16. Differences in outcome of PVL, embolization / migration 17.Assessment of PM dependency at 3 months post implant 18.Vascular access complication rate according to the "Hostile Score" 19. Changes in functional status from baseline to follow-up assessments at 30 days and 12 months (e.g., New York Heart Association (NYHA) functional classification, quality of life measure: Kansas City Cardiomyopathy Questionnaire (KCCQ)) 20. Rehospitalization (procedure-related or valve-related hospitalization, and other cardiovascular hospitalization) at 30 days and 12 months
Key Valve Academic Research Consortium (VARC) 3 event definitions | 30 days, 12 months and annually through 5 years
  21. Paravalvular leak (none/trace, mild, moderate or severe) at discharge, 30 days, 12 months and annually (when collected) through 5 years 22. Changes in echocardiographic parameters from baseline to follow-up at 30 days, 12 months and annually (when collected) through 5 years (e.g., mean effective orifice area, mean transvalvular gradient) 23. Aortic valve reintervention at 30 days, 12 months, and annually through 5 years 24. Prosthetic valve endocarditis at 12 months and annually through 5 years 25. Structural valve deterioration at 12 months and annually through 5 years 26. Non-structural valve dysfunction at 12 months and annually through 5 years 27. Successful coronary access as needed at 12 months and annually through 5 years 28. Clinically significant prosthetic valve thrombosis at 12 months and annually through 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Policlinico San Donato, San Donato Milanese, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-07-18): https://cdn.clinicaltrials.gov/large-docs/98/NCT07359898/Prot_SAP_000.pdf
  • Informed Consent Form (2025-07-22): https://cdn.clinicaltrials.gov/large-docs/98/NCT07359898/ICF_001.pdf